CLINICAL TRIAL: NCT00517621
Title: A Multicenter Prospective Phase II Study Evaluating Peripheral Neurotoxicity by Using FACT-GOG/NTX Questionnaire in Patients With Ovarian Cancer in Relapse Treated by Paclitaxel +/- EPO. Validation of a French Version of This Questionnaire
Brief Title: Use of FACT-GOG/NTX Questionnaire in Peripheral Neurotoxicity & Validation of a French Version of This Questionnaire
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: ARCAGY/ GINECO GROUP (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ETAMINE
Record Dates: First submitted 2007-08-16; First posted 2007-08-17 (Estimated); Last update posted 2011-02-25 (Estimated); Status verified 2011-02

CONDITIONS: Ovarian Cancer; Fallopian Tube Cancer; Peritoneal Neoplasms
Keywords: Peritoneal cancer; Relapse or progression
MeSH Terms: conditions — Ovarian Neoplasms; Fallopian Tube Neoplasms; Peritoneal Neoplasms; Recurrence; Disease Progression | interventions — Paclitaxel

INTERVENTIONS:
Drug: Paclitaxel
Drug: EPO

SUMMARY:
validation of a french version of FACT-GOG/NTX and using this questionnaire to evaluate the incidence of the peripheral neurotoxicity in patients treated for ovarian cancer with paclitaxel associated or not with EPO.

ELIGIBILITY:
Inclusion Criteria:

* Femal patient aged > 18 years
* Histologically proven diagnosis of cancer of the ovary, the fallopian tube or peritoneal
* patients whose disease progresses or relapses
* patients having received at least a line of platinum-based chemotherapy
* patients whose treatment of relapse is envisaged to comprise paclitaxel
* patients who will receive EPO for treatment of their anaemia
* ECOG performans status < 2
* life expectancy > 16 weeks
* patient who has clearly given her consent by signing on informed consent form prior to participation

Exclusion Criteria:

* peripheral neuropathy grade > 2
* history of ischemic cardiopathy, congestive heart failure (NYHA>2), arrhythmia, hypertension or significant valvulopathy
* abnormal biological values
* A therapy or a serious disease which could involve a risk for the patient or interfere with the aims of the study
* patient who is pregnant, breast feeding or using inadequate contraception
* concomitant therapy by a potentially neurotoxic drug
* concomitant inclusion in another therapeutic trial which could interfere with the aims of the study
* patient who for familial, sociological, geographical or psychological condition could not be followed correctly

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2006-02; Primary Completion 2010-09 (Actual); Study Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
Validation of a french version of FACT-GOG/NTX of peripheral neurotoxicity questionnaire

SECONDARY OUTCOMES:
- incidence and severity of the peripheral neurotoxicity according to whether the patients are treated or not by EPO
- variation of the rate of haemoglobin during chemotherapy
- Incidence of the thrombo-embolic events according to whether the patients are treated or not by EPO

CONTACTS AND LOCATIONS:
Overall Officials: Laure COPEL, Physician, Principal Investigator — Institut Curie Paris
Locations (1):
- HOTEL DIEU Hospital, Paris, France